CLINICAL TRIAL: NCT00785889
Title: A Randomized Controlled Comparison of Warm Water Infusion in Lieu of Air Insufflation vs. Air Insufflation for Aiding Colonoscopy Insertion in Sedated Patients Undergoing Colorectal Cancer (CRC) Screening and Surveillance.
Brief Title: RCT of Air Insufflation Versus Water Infusion Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Bay Institute for Research and Education (Other)
Responsible Party: Joseph Leung, M.D., GI Section, Northern California Health Care System
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: EBIRE-GI-001
Record Dates: First submitted 2008-11-03; First posted 2008-11-05 (Estimated); Last update posted 2008-11-14 (Estimated); Status verified 2008-11

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer screening; optical colonoscopy; water method; sedation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: water infusion colonoscopy — water infusion in lieu of air insufflation for screening colonoscopy
  Other Names: optical colonoscopy, water infusion colonoscopy

SUMMARY:
Compared with the conventional (air) method, patients examined by the study (water) method have lower pain scores and require less medication but have similar cecal intubation rate and willingness to repeat future colonoscopy.

DETAILED DESCRIPTION:
Background: A novel water method permitted 52% of patients accepting on-demand sedation to complete colonoscopy without medications and significantly increased successful cecal intubation from 76% to 97% in patients accepting scheduled unsedated colonoscopy.

Aim: To perform a randomized controlled trial comparing air insufflation (conventional method) vs. water infusion in lieu of air (study method) colonoscopy in minimally sedated patients.

Hypothesis: Compared with the conventional method, patients examined by the study method have lower pain scores and require less medication but have similar cecal intubation rate and willingness to repeat future colonoscopy.

Setting: Outpatient colonoscopy in a single VA hospital Methods: After informed consent and standard bowel preparation, patients received pre-medications administered as 0.5 increment of Fentanyl (25 μg) and 0.5 increment of Versed (1 mg) plus 50 mg Diphenhydramine. The conventional and the study method for colonoscopy were implemented as previously described. Additional pain medications were administered at the patients' request.

Outcome measures: Increments of medications, pain scores, cecal intubation and willingness to repeat colonoscopy.

Limitations: Single VA site, older male population

ELIGIBILITY:
Inclusion Criteria:

* healthy individual 50 years or older
* eligible for colorectal cancer screening or surveillance

Exclusion Criteria:

* patients who do not understand or failed to sign informed consent

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Increments of medications used for sedation | duration of procedure

SECONDARY OUTCOMES:
pain scores during colonoscopy | duration of procedure
success with cecal intubation | during procedure
willingness to repeat colonoscopy | after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Leung, MD, Principal Investigator — Sacramento VA Medical Center, GI Section
Locations (1):
- Sacramento VA Medical Center, VANCHCS, Mather, California, United States

REFERENCES:
- [Background] Leung JW, Mann S, Leung FW. Options for screening colonoscopy without sedation: a pilot study in United States veterans. Aliment Pharmacol Ther. 2007 Aug 15;26(4):627-31. doi: 10.1111/j.1365-2036.2007.03404.x. PMID 17661766
- [Background] Leung FW. Water-related techniques for performance of colonoscopy. Dig Dis Sci. 2008 Nov;53(11):2847-50. doi: 10.1007/s10620-008-0259-1. Epub 2008 May 7. PMID 18461455
- [Background] Leung FW, Aharonian HS, Guth PH, Chu SK, Nguyen BD, Simpson P. Involvement of trainees in routine unsedated colonoscopy: review of a pilot experience. Gastrointest Endosc. 2008 Apr;67(4):718-22. doi: 10.1016/j.gie.2007.11.040. PMID 18374030
- [Derived] Leung JW, Mann SK, Siao-Salera R, Ransibrahmanakul K, Lim B, Cabrera H, Canete W, Barredo P, Gutierrez R, Leung FW. A randomized, controlled comparison of warm water infusion in lieu of air insufflation versus air insufflation for aiding colonoscopy insertion in sedated patients undergoing colorectal cancer screening and surveillance. Gastrointest Endosc. 2009 Sep;70(3):505-10. doi: 10.1016/j.gie.2008.12.253. Epub 2009 Jun 24. PMID 19555938